CLINICAL TRIAL: NCT01236521
Title: Care Management for the Effective Use of Opioids (CAMEO)
Brief Title: Care Management for the Effective Use of Opioids
Acronym: CAMEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 10-128
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain; Pain
Keywords: Back pain; Care Management; Pain; Patient outcomes; Patient-center Care; Primary care
MeSH Terms: conditions — Low Back Pain; Pain; Back Pain | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Pharmacological (MED) (Experimental): Subjects in the Pharmacological (MED) arm will receive at least 8 contacts with the nurse care managers (NCM) over the trial period. Participants will have an initial visit at baseline to assess their current and past treatments for chronic lower back pain, pain intensity, and pain-related limitations. Patients' opioids will be adjusted and/or co-analgesics (or adjuvants) will be initiated. During follow-up calls, patients' pain severity, response to treatment, adherence, adverse effects, and desire to change current treatment will be assessed. Follow-up NCM telephone contacts will occur at 2 and 4 weeks after baseline, and months 2, 3, 4, 6, and 9 months. On average, these calls last between 10 to 20 minutes. Detailed logs will be kept of the timing and content of patient contacts.
  Interventions: Drug: Pharmacological (MED)
- Arm 2: Behavioral treatment (CBT) (Experimental): Veterans randomized to behavioral treatment arm (CBT) will receive a series of 8 pain self-management/coping skills training sessions delivered by one of three primary-care based clinical psychologists. Since optimal application of non-pharmacological interventions for pain involves tailoring to patient needs, participants will be introduced to a menu of self-management and coping skills rather than receive a prescribed program. Delivery of the behavioral intervention will employ a flexible approach that is easily adapted to individual preferences and perceived need for learning specific pain coping skills. Tailoring will include the selection of relevant content and skills and assessment of readiness to change behaviors.
  Interventions: Behavioral: Behavioral treatment (CBT)

INTERVENTIONS:
Drug: Pharmacological (MED) — During the baseline assessment, the nurse care managers will determine current and past treatments for chronic lower back pain and establish whether or not patients have had an adequate trial (i.e., were analgesics sufficiently dosed). If not, the nurse care manager in conjunction with study doctors will recommend an adjustment of the patients' opioid or initiate treatment with a co-analgesic with appropriate dosing and scheduling.
  The Patients in the MED arm will be asked to sign an opioid treatment agreement at enrollment.
  Other Names: Co-analgesic algorithm
  Arms: Arm 1: Pharmacological (MED)
Behavioral: Behavioral treatment (CBT) — There will be 8 sessions of pain self-management and coping skills.
  Other Names: Pain self-management/coping skills treatment
  Arms: Arm 2: Behavioral treatment (CBT)

SUMMARY:
The CAre Management for the Effective use of Opioids (CAMEO) trial is a 2-arm randomized clinical trial to compare the effectiveness of pharmacological vs. behavioral approaches for chronic lower back pain. The study aims are to compare the interventions' (PHARM vs. BEH) effects on pain intensity, pain interference, function, and other pain relevant outcomes over 12 months.

DETAILED DESCRIPTION:
The general purpose of the CAre Management for the Effective use of Opioids (CAMEO) study is to develop, test, and implement novel treatments and care delivery models that address barriers to effective pain management and that can be practicably applied in VA primary care settings for chronic low back pain (CLBP). The CAMEO trial is a 2-arm randomized clinical trial to compare the effectiveness of pharmacological vs. behavioral approaches for CLBP.

The investigators' study sample will target 272 Veterans with moderate to severe CLBP despite long-term opioid therapy. Patients from five primary care clinics at the Roudebush VA Medical Center and two community based outpatient clinics will be recruited to participate in CAMEO and randomized to one of two treatment arms. The pharmacological arm will involve guideline-concordant opioid management coupled with algorithm-based co-analgesic treatment (MED). Patients in the behavioral arm (CBT) will receive pain self-management/coping skills training. The trial will last 12-months and all participants will undergo comprehensive outcome assessments at baseline, 3, 6, 9, and 12 months.

Study Aims: Among Veterans with chronic low back pain refractory to long-term opioid therapy

1. To compare the interventions' (MED vs. CBT) effects on pain intensity and function over 12 months
2. To compare the interventions' effects (MED vs. CBT) on other relevant outcomes

   * Health-related quality of life
   * Pain Catastrophizing
   * Depression
   * Anxiety
   * Disability
   * Opioid misuse and opioid dose

ELIGIBILITY:
Inclusion Criteria:

Veterans will be eligible if they have:

* chronic lower back pain of at least moderate intensity
* pain for 6 months
* on chronic opioid therapy
* and access to a working telephone

Exclusion Criteria:

Exclusion criteria includes:

* severe medical conditions
* active psychosis
* schizophrenia
* active suicidal ideation
* pending back surgery
* moderately severe cognitive impairment
* involvement in ongoing pain trials
* and pregnant or trying to become pregnant

The investigators will exclude Veterans with an active substance use disorder (i.e., those currently in treatment), but to maximize generalizability the investigators will not exclude those with a past history of substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Bair, MD MS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Upon request, we will share data with other researchers

REFERENCES:
- [Result] Chen CX, Kroenke K, Stump TE, Kean J, Carpenter JS, Krebs EE, Bair MJ, Damush TM, Monahan PO. Estimating minimally important differences for the PROMIS pain interference scales: results from 3 randomized clinical trials. Pain. 2018 Apr;159(4):775-782. doi: 10.1097/j.pain.0000000000001121. PMID 29200181
- [Result] Chen CX, Kroenke K, Stump T, Kean J, Krebs EE, Bair MJ, Damush T, Monahan PO. Comparative Responsiveness of the PROMIS Pain Interference Short Forms With Legacy Pain Measures: Results From Three Randomized Clinical Trials. J Pain. 2019 Jun;20(6):664-675. doi: 10.1016/j.jpain.2018.11.010. Epub 2018 Dec 6. PMID 30529442
- [Result] Bair MJ, Outcalt SD, Slaven JE, Kroenke K, Kempf C, Zillich AJ, Damush TM, Saha C, French DD, Krebs EE. Care Management for the Effective Use of Opioids (CAMEO): A Randomized Trial. Abstracts of the 77th Annual Scientific Meeting, March 6-9, 2019. Vancouver, BC, Canada. Abstract 1734. [Abstract]. Psychosomatic medicine. 2019 May 1; 81(4):A-149.
- [Result] Kroenke K, Stump TE, Chen CX, Kean J, Bair MJ, Damush TM, Krebs EE, Monahan PO. Minimally important differences and severity thresholds are estimated for the PROMIS depression scales from three randomized clinical trials. J Affect Disord. 2020 Apr 1;266:100-108. doi: 10.1016/j.jad.2020.01.101. Epub 2020 Jan 23. PMID 32056864
- [Result] Kroenke K, Stump TE, Chen CX, Kean J, Damush TM, Bair MJ, Krebs EE, Monahan PO. Responsiveness of PROMIS and Patient Health Questionnaire (PHQ) Depression Scales in three clinical trials. Health Qual Life Outcomes. 2021 Feb 4;19(1):41. doi: 10.1186/s12955-021-01674-3. PMID 33541362
- [Result] Kroenke K, Stump TE, Kean J, Krebs EE, Damush TM, Bair MJ, Monahan PO. Diagnostic operating characteristics of PROMIS scales in screening for depression. J Psychosom Res. 2021 Aug;147:110532. doi: 10.1016/j.jpsychores.2021.110532. Epub 2021 May 25. PMID 34052655
- [Result] Bushey MA, Slaven J, Outcalt SD, Kroenke K, Kempf C, Froman A, Sargent C, Baecher B, Zillich A, Damush TM, Saha C, French DD, Bair MJ. Design and methods of the Care Management for the Effective Use of Opioids (CAMEO) trial. Contemp Clin Trials. 2021 Jul;106:106456. doi: 10.1016/j.cct.2021.106456. Epub 2021 May 25. PMID 34048943
- [Result] Bushey MA, Slaven JE, Outcalt SD, Kroenke K, Kempf C, Froman A, Sargent C, Baecher B, Zillich AJ, Damush TM, Saha C, French DD, Bair MJ. Effect of Medication Optimization vs Cognitive Behavioral Therapy Among US Veterans With Chronic Low Back Pain Receiving Long-term Opioid Therapy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242533. doi: 10.1001/jamanetworkopen.2022.42533. PMID 36394874
- [Result] Midboe AM, Lewis ET, Paik MC, Gallagher RM, Rosenberg JM, Goodman F, Kerns RD, Becker WC, Trafton JA. Measurement of adherence to clinical practice guidelines for opioid therapy for chronic pain. Transl Behav Med. 2012 Mar;2(1):57-64. doi: 10.1007/s13142-011-0104-5. PMID 24073098
- [Derived] Koechlin H, Locher C, Barke A, Korwisi B. Retrospective identification of the diagnosis of chronic primary musculoskeletal pain: a pragmatic suggestion by The Pain Net. Pain. 2025 Feb 1;166(2):311-314. doi: 10.1097/j.pain.0000000000003380. Epub 2024 Sep 3. No abstract available. PMID 39172815

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pharmacological (PHARM): Subjects in the Pharmacological (PHARM) arm received at least 8 contacts with the nurse care managers (NCM) over the trial period. Participants had an initial visit at baseline to assess their current and past treatments for chronic lower back pain, pain intensity, and pain-related limitations. During follow-up calls, patients' pain severity, response to treatment, adherence, adverse effects, and desire to change current treatment was assessed.
  Analgesic and co-analgesic therapy: During the baseline assessment, the nurse care managers determined current and past treatments for chronic lower back pain.
- Arm 2: Behavioral Treatment (BEH): Veterans randomized to behavioral treatment arm (BEH) received a series of 8 pain self-management/coping skills training sessions delivered by one of three primary-care based clinical psychologists.
Period: Overall Study
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Started | 131 | 130
3-month Completed | 122 | 118
6-month Completed | 121 | 114
9-month Completed | 105 | 98
12-moth Completed | 108 | 105
Completed | 108 | 105
Not Completed | 23 | 25
Not completed — Withdrawal by Subject | 12 | 17
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Pharmacological (PHARM): Subjects in the Pharmacological (PHARM) arm will receive at least 8 contacts with the nurse care managers (NCM) over the trial period. During follow-up calls, patients' pain severity, response to treatment, adherence, adverse effects, and desire to change current treatment will be assessed. During the baseline assessment, the nurse care managers will determine current and past treatments for chronic lower back pain and establish whether or not patients have had an adequate trial (i.e., were analgesics sufficiently dosed). If not, the nurse care manager in conjunction with study doctors will recommend an adjustment of the patients' opioid or initiate treatment with a co-analgesic with appropriate dosing and scheduling.
- Arm 2: Behavioral Treatment (BEH): Veterans randomized to behavioral treatment arm (BEH) will receive a series of 8 pain self-management/coping skills training sessions delivered by one of three primary-care based clinical psychologists.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH) | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.8) | 58.2 (9.2) | 57.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 124 | 117 | 241
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 25 | 54
  White | 91 | 100 | 191
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Total Score at Baseline and Change Score From Baseline at 3, 6, 9, and 12 Months
Description: The Brief Pain Inventory Total Score combines scores from the BPI Pain Intensity subscale and the BPI Pain Interference subscale. This scale provides a total score from 0 (no pain/no pain interference) to 10 (worst pain imaginable/completely interferes). We report below the baseline score on the 0 to 10 scale. At each follow-up time point (3, 6, 9, and 12 months) we report the change from baseline to follow-up. This value was calculated as the baseline score minus the follow-up score.
Time Frame: Baseline and 3, 6, 9, and 12 months
Population: We analyzed those participants with available data. We had more participants at baseline than the follow-up time points at 3, 6, 9, and 12 months due to attrition and no available data among those who dropped out of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Pharmacological (PHARM): Subjects in the Pharmacological (PHARM) arm received at least 8 contacts with the nurse care managers (NCM) over the trial period.
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
units on a scale
  Baseline | 6.45 (1.79) | 6.49 (1.67)
  3 months: number analyzed (Participants) | 121 | 118
  3 months | 5.41 (2.10) | 5.86 (1.91)
  6 months: number analyzed (Participants) | 121 | 114
  6 months | 5.39 (2.21) | 5.85 (1.84)
  9 months: number analyzed (Participants) | 105 | 98
  9 months | 5.29 (2.25) | 5.66 (1.91)
  12 months: number analyzed (Participants) | 108 | 105
  12 months | 5.31 (2.27) | 5.85 (1.98)
Statistical Analysis 1: Comparison: Arm 1: Pharmacological (PHARM) vs Arm 2: Behavioral Treatment (BEH); Test type: Superiority; p = 0.0385, Mixed Models Analysis; Mean Difference (Net) = 0.39, Standard Deviation 0.13

2. Primary Outcome: Brief Pain Inventory Pain Intensity Score at Baseline and Each Follow-up Time Point
Description: The Brief Pain Inventory pain intensity score is scored from 0 (no pain) to 10 (worst pain imaginable). We report below the baseline score on the 0 to 10 scale. At each follow-up time point (3, 6, 9, and 12 months) we report the change from baseline to follow-up. This value was calculated as the baseline score minus the follow-up score.
Time Frame: Baseline and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
units on a scale
  Baseline | 6.78 (1.65) | 6.76 (1.47)
  3 months: number analyzed (Participants) | 121 | 118
  3 months | 5.96 (1.86) | 6.24 (1.56)
  6 months: number analyzed (Participants) | 121 | 114
  6 months | 5.94 (1.95) | 6.45 (1.60)
  9 months: number analyzed (Participants) | 105 | 98
  9 months | 5.84 (1.83) | 6.18 (1.69)
  12 months: number analyzed (Participants) | 108 | 105
  12 months | 5.76 (2.14) | 6.36 (1.59)
Statistical Analysis 1: Comparison: Arm 1: Pharmacological (PHARM) vs Arm 2: Behavioral Treatment (BEH); Test type: Superiority; p = 0.0067, Mixed Models Analysis; Mean Difference (Net) = 0.44, Standard Deviation 0.11

3. Primary Outcome: Brief Pain Inventory Pain Interference Scale Score
Description: The Brief Pain Inventory Pain Interference Scale score assesses if pain interferes with 7 common activities. This scale is score 0 (no interference) to 10 (high interference). The 7-items are averaged to give a score.
Time Frame: Baseline and 3, 6, 9, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 6.34 (2.07) | 6.39 (1.99)
  3 months: number analyzed (Participants) | 121 | 118
  3 months | 5.19 (2.38) | 5.71 (2.28)
  6 months: number analyzed (Participants) | 121 | 114
  6 months | 5.17 (2.51) | 5.61 (2.15)
  9 months: number analyzed (Participants) | 105 | 98
  9 months | 5.08 (2.57) | 5.47 (2.19)
  12 months: number analyzed (Participants) | 108 | 105
  12 months | 5.15 (2.46) | 5.68 (2.30)
Statistical Analysis 1: Comparison: Arm 1: Pharmacological (PHARM) vs Arm 2: Behavioral Treatment (BEH); Test type: Superiority; p = 0.0740, Mixed Models Analysis; Median Difference (Net) = 0.39, Standard Deviation 0.15

4. Secondary Outcome: Pain Catastrophizing Scale
Description: The Pain Catastrophizing Scale a 13-item scale that assesses catastrophizing - a pain belief that have been found to be strong predictor of poor treatment response. It is scored from 0 (no catastrophizing) to 52 (severe catastrophizing)
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 23.95 (12.77) | 24.44 (11.27)
  6 months | 21.64 (13.20) | 20.41 (12.54)
  12 months | 22.14 (13.84) | 20.43 (12.04)

5. Secondary Outcome: Roland Morris Disability Scale
Description: The Roland Morris Disability Scale is a 24-item pain-specific measure of physical disability. It provides a score from 0 (no disability) to 24 (high disability)
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 16.59 (4.70) | 16.72 (4.15)
  3 months | 15.55 (5.18) | 15.80 (5.20)
  6 months | 15.32 (5.20) | 15.34 (5.50)
  9 months | 15.54 (5.53) | 15.33 (5.50)
  12 months | 15.60 (5.85) | 16.58 (5.34)

6. Secondary Outcome: Patient Health Questionnaire-9
Description: The Patient Health Questionnaire-9 is used to assess depression severity. It's 9-items that are scored from 0 (no depression) to 27 (severe depression)
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 11.18 (6.40) | 11.19 (5.82)
  3 months | 9.74 (6.33) | 9.94 (6.14)
  6 months | 9.74 (6.56) | 10.04 (6.12)
  9 months | 9.67 (6.41) | 9.84 (5.68)
  12 months | 10.13 (6.95) | 10.53 (6.21)

7. Secondary Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: The GAD-7 is a measure of anxiety. The GAD-7 consists of 7 items that are scored from 0 (no anxiety) to 21 (severe anxiety)
Time Frame: Baseline, 3 months, 6 months, 9 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 6.68 (5.13) | 6.81 (4.63)
  3 months | 6.65 (4.50) | 6.08 (4.57)
  6 months | 6.00 (5.23) | 6.22 (4.88)
  9 months | 6.30 (4.92) | 5.92 (4.83)
  12 months | 6.41 (5.30) | 7.02 (4.98)

8. Secondary Outcome: AUDIT-C
Description: The AUDIT-C is validated as an effective screening test and diagnostic tool for alcohol misuse in primary care samples. It is scored on 0 to 10 score with higher scores representing alcohol misuse
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 5.65 (5.51) | 5.87 (5.71)
  6 months | 5.42 (5.69) | 5.75 (5.40)
  12 months | 5.06 (5.58) | 5.36 (5.66)

9. Secondary Outcome: Current Opioid Misuse Measure (COMM)
Description: The COMM (Current Opioid Misuse Measure) is a 17-item instrument designed to monitor misuse and aberrant behaviors in patients prescribed opioids. The scale is scored from 0 (no evidence of opioid misuse or aberrant behaviors) to 64 (strong evidence for opioid misuse and aberrant behaviors)
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 8.73 (6.81) | 8.87 (6.54)
  6 months | 7.29 (6.96) | 8.20 (6.85)
  12 months | 7.60 (6.96) | 8.96 (7.94)

10. Secondary Outcome: SF-36 General Health Perception
Description: The SF-36 is a subscale that assesses the self-reported general health. It is scored on a 0 to 100 scale with higher scores representing greater perceived general health
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 43.66 (20.92) | 45.39 (18.64)
  6 months | 45.85 (19.89) | 45.83 (20.40)
  12 months | 42.70 (23.03) | 42.44 (20.17)

11. Secondary Outcome: SF-36 Vitality Scale
Description: The SF-36 vital score is a subscale that assesses participants' vitality/energy. It is scored on a 0 to 100 scale with higher scores representing greater vitality/energy.
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 38.64 (16.98) | 35.08 (16.17)
  6 months | 40.00 (17.50) | 38.33 (17.06)
  12 months | 40.51 (16.28) | 38.19 (15.74)

12. Secondary Outcome: SF-36 Social Functioning Scale
Description: The SF-36 social functioning scale is a subscale that assesses the self-reported social functioning. It is scored on a 0 to 100 scale with higher scores representing better social functioning.
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
Number analyzed (Participants) | 131 | 130
scores on a scale
  Baseline | 48.47 (27.21) | 49.81 (29.32)
  6 months | 55.79 (29.67) | 51.10 (27.40)
  12 months | 55.72 (28.49) | 52.02 (28.12)

ADVERSE EVENTS:
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Groups:
- Arm 1: Pharmacological (PHARM): Nurse care managers followed an analgesic algorithm; supervised by study physicians
- Arm 2: Behavioral Treatment (BEH): Clinical psychologist delivered pain self-management/pain coping skills to Veterans
Arm/Group | Arm 1: Pharmacological (PHARM) | Arm 2: Behavioral Treatment (BEH)
All-Cause Mortality (participants affected / at risk) | 2/131 | 1/130
Serious Adverse Events (participants affected / at risk) | 6/131 | 1/130
Other Adverse Events (participants affected / at risk) | 10/131 | 2/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pharmacological (PHARM) (N=131) | Arm 2: Behavioral Treatment (BEH) (N=130)
Knee Replacement Surgery (Surgical and medical procedures) | 1 (1) | 1 (1) — Patient was admitted for knee replacement surgery
Small Bowel Obstruction (Gastrointestinal disorders) | 2 (6) | 0 (0) — Participant was admitted to hospital for small bowel obstruction Another participant was admitted for dehydration due to high output ileostomy
Urinary Tract Infection and Sepsis (Infections and infestations) | 2 (2) | 0 (0) — Participant was admitted for urinary tract infection and sepsis Another participant was admitted with fever and cough. Discharge diagnosis was viral illness
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Participant admitted for atrial fibrillation with rapid ventricular rate
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pharmacological (PHARM) (N=131) | Arm 2: Behavioral Treatment (BEH) (N=130)
other adverse event (Infections and infestations) | 6 (6) | 0 (0)
other adverse event (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
other adverse event (Cardiac disorders) | 1 (2) | 0 (0)
other adverse event (Gastrointestinal disorders) | 2 (4) | 0 (0)
other adverse event (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes